CLINICAL TRIAL: NCT04531917
Title: The Effect of Pain Neuroscience Education and Behavioural Graded Activity Compared to Usual Care on Chronic Pain in Breast Cancer Survivors: a Randomised Controlled Trial
Brief Title: The Effect of Pain Neuroscience Education and Behavioural Graded Activity on Chronic Pain in Breast Cancer Survivors
Acronym: BCS-PAIN
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitair Ziekenhuis Brussel (Other)
Collaborators: Fund for Scientific Research, Flanders, Belgium (Other); Vrije Universiteit Brussel (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 11B1920N_BCS-PAIN
Record Dates: First submitted 2020-08-18; First posted 2020-08-31 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Breast Neoplasms; Survivors; Chronic Pain
Keywords: Behavioural Graded Activity; Pain Neuroscience Education
MeSH Terms: conditions — Breast Neoplasms; Chronic Pain

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pain Neuroscience Education + Behavioural Graded Activity (Experimental): Patients allocated to the intervention group will receive a 12-week treatment program that consists of 6 sessions, in which 'Pain Neuroscience Education' and 'Behavioural Graded Activity' will be integrated.
  Interventions: Other: Pain Neuroscience Education; Other: Behavioural Graded Activity
- Usual care (Active Comparator): Patients allocated to the control group will receive an information leaflet from "Kom op tegen kanker" regarding "Pain in and after cancer".
  Interventions: Other: Usual care

INTERVENTIONS:
Other: Pain Neuroscience Education — Pain Neuroscience Education (PNE) teaches patients about complex pain mechanisms known to be of importance in pain following breast cancer such as malfunctioning of the endogenous analgesic system and pain memories.
  Arms: Pain Neuroscience Education + Behavioural Graded Activity
Other: Behavioural Graded Activity — Patients in the experimental group will receive a behavioural treatment integrated within the concepts of operant conditioning. The purpose of Behavioural Graded Activity (BGA) is to increase the level of physical activity in the patient's daily lives in a time-contingent manner. On top of that, a healthy behaviour will be positively reinforced to consequently create a withdrawal of the attention towards pain behaviour, which is seen as an unreliable "alarm sign" in chronic pain patients. The implementation of BGA after PNE is described in the guideline reported by the International Association for the Study of Pain.
  Arms: Pain Neuroscience Education + Behavioural Graded Activity
Other: Usual care — The content of the leaflet has a biomedical approach in explaining pain and providing information on the different pain medication classes. This leaflet is mostly available in waiting rooms of oncology centres and units of the Flemish part of Belgium.
  Arms: Usual care

SUMMARY:
Chronic pain in breast cancer survivors (BCS) is of considerable concern as it impacts the health-related quality of life (HRQoL) and activities of daily living negatively. Over the past decades, awareness has raised the value of pain neuroscience education (PNE) in chronic pain. However, pain education remains underused in oncology and is often restricted to a biomedical management, which falls short in explaining persistent pain following cancer. Since PNE alone has rather small effect sizes, it should ideally be combined with a physical part, 'behavioural graded activity' (BGA). Therefore, the purpose of this study is to investigate the effectiveness of PNE with BGA compared to usual care on chronic pain in BCS.

A multi-centre, parallel, two-arm, double-blinded superiority with a three months intervention and two years follow-up will be conducted in 200 BCS with chronic pain. These will be randomly assigned to the intervention or usual care group. The intervention group will receive 6 sessions, in which PNE and BGA will be integrated. Whereas, the usual care group will receive an information leaflet regarding "Pain in and after cancer".

The primary objective of the present study is to examine whether the combination of PNE and BGA has an added value in decreasing the pain intensity compared to the usual care in BCS with chronic pain. The secondary objectives are to investigate whether the combination of PNE and BGA has the ability to reduce endogenous hyperalgesia and improve HRQoL compared to the usual care in BCS with chronic pain.

ELIGIBILITY:
Inclusion Criteria:

* To meet the definition introduced by the National Cancer Institute's Office of Cancer Survivorship, in which a cancer survivor is a patient with a history of cancer that is beyond the acute diagnosis and treatment phase. Patients need to be cancer-free and should have finished their primary treatment with a curative intent for at least 3 months prior to study participation. Adjuvant hormonal therapy and immunotherapy form the exception to the rule and are tolerated.
* To report a pain severity of at least 3 out of 10 on pain visual analogue scale.
* To be able to speak and read in Dutch in order to give informed consent and to complete the assessment tools. Written and signed consent will be obtained from all participants.

Exclusion Criteria:

* Suffering from dementia or cognitive impairment (unable to understand the test instructions and/or Mini Mental State Examination score <23/30).
* Suffering from severe psychological or psychiatric diseases.
* Diagnosis of new neoplasms or metastases.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2020-10-12 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change in pain intensity and pain interference | T1: baseline (within one week before randomisation) and T3: 3 months after intervention (w 26)
  Change between baseline (T1) and 3 months post-intervention (T3)
  * Measured with the 'Brief Pain Inventory'
  * The minimum and maximum values: 0, 10
  * Higher score means a worse outcome
Self-reported pain intensity and pain interference | T1: baseline (within one week before randomisation)
  * Measured with the 'Brief Pain Inventory'
  * The minimum and maximum values: 0, 10
  * Higher score means a worse outcome
Self-reported pain intensity and pain interference | T2: after finishing intervention (week 13)
  * Measured with the 'Brief Pain Inventory'
  * The minimum and maximum values: 0, 10
  * Higher score means a worse outcome
Self-reported pain intensity and pain interference | T3: 3 months after intervention (week 26)
  * Measured with the 'Brief Pain Inventory'
  * The minimum and maximum values: 0, 10
  * Higher score means a worse outcome
Self-reported pain intensity and pain interference | T4: 1 year after intervention (week 64)
  * Measured with the 'Brief Pain Inventory'
  * The minimum and maximum values: 0, 10
  * Higher score means a worse outcome
Self-reported pain intensity and pain interference | T5: 2 years after intervention (week 116)
  * Measured with the 'Brief Pain Inventory'
  * The minimum and maximum values: 0, 10
  * Higher score means a worse outcome

SECONDARY OUTCOMES:
Self-reported health-related quality of life | T1: baseline (within one week before randomisation), T2: after finishing intervention (w 13), T3: 3 months after intervention (w 26), T4: 1 year after intervention (w 64) and T5: 2 years after intervention (w 116)
  * Measured with the 'European Organisation for Research and Treatment of Cancer Core Quality of Life Questionnaire (EORTC-QLQ-C30)'
  * The minimum and maximum values: 0, 100
  * Higher score means a better outcome
Temperature detection threshold | T1: baseline (within one week before randomisation), T2: after finishing intervention (w 13) and T3: 3 months after intervention (w 26)
  Assessed by the Medoc TSA-II Neurosensory Analyzer.
Pain detection threshold | T1: baseline (within one week before randomisation), T2: after finishing intervention (w 13) and T3: 3 months after intervention (w 26)
  Assessed by the digital algometer, the Medoc TSA-II Neurosensory Analyzer and a manual blood pressure cuff.
Pain tolerance threshold | T1: baseline (within one week before randomisation), T2: after finishing intervention (w 13) and T3: 3 months after intervention (w 26)
  Assessed by a manual blood pressure cuff.
Endogenous pain inhibition | T1: baseline (within one week before randomisation), T2: after finishing intervention (w 13) and T3: 3 months after intervention (w 26)
  Assessed objectively by conditioned pain modulation paradigm. A manual blood pressure is the conditioned stimulus, and the digital algometer and the Medoc TSA-II Neurosensory Analyzer are testing stimuli.
Endogenous pain facilitation | T1: baseline (within one week before randomisation), T2: after finishing intervention (w 13) and T3: 3 months after intervention (w 26)
  Assessed objectively by temporal summation paradigm. Ten testing stimuli will be applied, and subjects will be asked to rate their pain intensity on the first, fifth and tenth stimulus by using the Visual Analogue Scale.

OTHER OUTCOMES:
Self-reported pain | T1: baseline (within one week before randomisation), T2: after finishing intervention (w 13), T3: 3 months after intervention (w 26), T4: 1 year after intervention (w 64) and T5: 2 years after intervention (w 116)
  * Measured with the 'Visual Analogue Scale'
  * The minimum and maximum values: 0mm, 100mm
  * Higher score means a worse outcome
Self-reported neuropathic pain | T1: baseline (within one week before randomisation), T2: after finishing intervention (w 13), T3: 3 months after intervention (w 26), T4: 1 year after intervention (w 64) and T5: 2 years after intervention (w 116)
  * Measured with the 'Douleur Neuropatique 4'
  * The minimum and maximum values: 0, 10
  * Higher score means a worse outcome
  * A score of 4 or higher indicates neuropathic pain
Self-reported central sensitization | T1: baseline (within one week before randomisation), T2: after finishing intervention (w 13), T3: 3 months after intervention (w 26), T4: 1 year after intervention (w 64) and T5: 2 years after intervention (w 116)
  * Measured with the 'Central Sensitization Index'
  * The minimum and maximum values: 0, 100
  * Higher score means a worse outcome
  * A score of 40 or higher indicates the presence of central sensitization
Self-reported physical activity level | T1: baseline (within one week before randomisation), T2: after finishing intervention (w 13), T3: 3 months after intervention (w 26), T4: 1 year after intervention (w 64) and T5: 2 years after intervention (w 116)
  * Measured with the 'International Physical Activity Questionnaire short form'
  * Total physical activity in MET-min/week and time spent sitting
Self-reported physical activity level | During the intervention and T2: after finishing intervention (w 13)
  * Measured with the 'logbook'
  * Subjects enrolled in the intervention arm will have to fill in the logbook on daily basis.
Self-reported sleep quality | T1: baseline (within one week before randomisation), T2: after finishing intervention (w 13), T3: 3 months after intervention (w 26), T4: 1 year after intervention (w 64) and T5: 2 years after intervention (w 116)
  * Measured with the 'Pittsburgh Sleep Quality Index'
  * The minimum and maximum values: 0, 21
  * Higher score means a worse outcome
  * A scores above 5 indicates poor global sleep quality
Self-reported insomnia severity | T1: baseline (within one week before randomisation), T2: after finishing intervention (w 13), T3: 3 months after intervention (w 26), T4: 1 year after intervention (w 64) and T5: 2 years after intervention (w 116)
  * Measured with the 'Insomnia Severity Index'
  * The minimum and maximum values: 0, 28
  * Higher score means a worse outcome
  * A scores of 8 or higher indicates insomnia
Self-reported fatigue | T1: baseline (within one week before randomisation), T2: after finishing intervention (w 13), T3: 3 months after intervention (w 26), T4: 1 year after intervention (w 64) and T5: 2 years after intervention (w 116)
  * Measured with the 'Fatigue Severity Scale'
  * The minimum and maximum values: 9, 63
  * Higher score means a worse outcome
Self-reported pain cognitions (pain catastrophizing) | T1: baseline (within one week before randomisation), T2: after finishing intervention (w 13), T3: 3 months after intervention (w 26), T4: 1 year after intervention (w 64) and T5: 2 years after intervention (w 116)
  * Measured with the 'Pain Catastrophizing Scale'
  * The minimum and maximum values: 0, 52
  * Higher score means a worse outcome
  * A scores of 30 or higher indicates pain catastrophizing thoughts
Self-reported pain cognitions (perceived injustice) | T1: baseline (within one week before randomisation), T2: after finishing intervention (w 13), T3: 3 months after intervention (w 26), T4: 1 year after intervention (w 64) and T5: 2 years after intervention (w 116)
  * Measured with the 'Injustice Experience Questionnaire'
  * The minimum and maximum values: 0, 48
  * Higher score means a worse outcome
Self-reported pain cognitions (illness perception) | T1: baseline (within one week before randomisation), T2: after finishing intervention (w 13), T3: 3 months after intervention (w 26), T4: 1 year after intervention (w 64) and T5: 2 years after intervention (w 116)
  * Measured with the 'the Brief Illness Perception Questionnaire'
  * The minimum and maximum values: 0, 10
  * Higher score means a worse outcome
Self-reported pain cognitions (pain vigilance and awareness) | T1: baseline (within one week before randomisation), T2: after finishing intervention (w 13), T3: 3 months after intervention (w 26), T4: 1 year after intervention (w 64) and T5: 2 years after intervention (w 116)
  * Measured with the 'Pain Vigilance and Awareness questionnaire'
  * The minimum and maximum values: 0, 90
  * Higher score means a worse outcome
Self-reported depression | T1: baseline (within one week before randomisation), T2: after finishing intervention (w 13), T3: 3 months after intervention (w 26), T4: 1 year after intervention (w 64) and T5: 2 years after intervention (w 116)
  * Measured with the 'Depression, Anxiety, Stress Scale'
  * The minimum and maximum values: 0, 21
  * Higher score means a worse outcome
Self-reported anxiety | T1: baseline (within one week before randomisation), T2: after finishing intervention (w 13), T3: 3 months after intervention (w 26), T4: 1 year after intervention (w 64) and T5: 2 years after intervention (w 116)
  * Measured with the 'Depression, Anxiety, Stress Scale'
  * The minimum and maximum values: 0, 21
  * Higher score means a worse outcome
Self-reported stress | T1: baseline (within one week before randomisation), T2: after finishing intervention (w 13), T3: 3 months after intervention (w 26), T4: 1 year after intervention (w 64) and T5: 2 years after intervention (w 116)
  * Measured with the 'Depression, Anxiety, Stress Scale'
  * The minimum and maximum values: 0, 21
  * Higher score means a worse outcome
Treatment adherence | During the intervention and T2: after finishing intervention (w 13)
  Patient adherence for the treatment sessions will be calculated as the ratio of the number of treatment sessions that were actually carried out versus the number of prescribed sessions.
Treatment compliance | During the intervention and T2: after finishing intervention (w 13)
  Compliance will be calculated as the ratio of the total training duration (recorded in the logbooks) versus the prescribed total training duration, multiplied by 100.
The presence of axillary web syndrome | T1: baseline (within one week before randomisation)
  The diagnosis of Axillary Web Syndrome (AWS) will be made clinically.
  * Scored on 5-point Likert scale (totally disagree, disagree, don't disagree/agree, agree, totally agree)
  * The presence of rope-like cords in the axilla to the wrist is assessed by inspection and/or palpation.
The presence of lymphedema | T1: baseline (within one week before randomisation)
  Lymphedema will be clinically diagnosed:
  The Stemmer sign is positive if the assessor is unable to pinch (between his/her thumb and index finger) the dorsal skin of proximal phalanx (second or third finger). A positive test confirms the presence of primary and secondary lymphedema of the arm(s).
  Single circumference measurement will only be performed if unilateral lymphedema is suspected. The arm circumference will be measured by a nylon tape measure with an accuracy of 1mm. The tape measure will be placed around the arm without tightening the tape at 30cm above the styloid process. Lymphedema is present if there is at least a difference of 10% between both arms.
The presence of arthralgia | T1: baseline (within one week before randomisation)
  To assess arthralgia the assessor will ask the patient two questions: "Do you experience symmetrical pain in the left and right shoulders, elbows, wrists, fingers, hips, knees, ankles and/or toes?" and "Do you experience morning stiffness? And if so, for how many minutes?"
Detection of inflammation or adhesion of the scar tissue | T1: baseline (within one week before randomisation)
  The scar tissue will be clinically scored. First, the assessor will inspect the affected (and painful) region for possible skin damage and will be looking for: wound disruption, hematoma (bruising), abscess (cavity filled with pus) and seroma (cavity filled with transparent liquid). Second, the he will inspect the presence of a possible inflammation process of the scar tissue and will be looking for signs such as: warmth, redness, etc. Third, he will assess the mobility of the scar. During this manual test, will be assessed whether the scar is moving relative to the underlying layers, which will be scored on a 5-point Likert scale with response possibilities: (totally disagree, disagree, don't disagree/agree, agree, totally agree).
Self-reported health care cost | T1: baseline (within one week before randomisation), T2: after finishing intervention (w 13), T3: 3 months after intervention (w 26), T4: 1 year after intervention (w 64) and T5: 2 years after intervention (w 116)
  * Measured with the 'Medical Consumption Questionnaire'
  * 38 questions to quantify the direct medical costs of a patients' total medical consumption, encompassing additional diagnostics, consultations, surgery including stay in hospitals, physiotherapy, medication and aids prescribed by the general practitioner as well as medication and aids purchased by the patients themselves.
Self-reported work absenteeism and productivity loss at work | T1: baseline (within one week before randomisation), T2: after finishing intervention (w 13), T3: 3 months after intervention (w 26), T4: 1 year after intervention (w 64) and T5: 2 years after intervention (w 116)
  * Measured with the 'Productivity Cost Questionnaire'
  * 20 questions to quantify the indirect costs outside health care but related to the disease (e.g. the costs due to absence of work and possible decreased productivity losses of paid and unpaid work).
Self-reported overall health status | T1: baseline (within one week before randomisation), T2: after finishing intervention (w 13), T3: 3 months after intervention (w 26), T4: 1 year after intervention (w 64) and T5: 2 years after intervention (w 116)
  * Measured with the 'EuroQol 5D instrument (EQ-5D-5L)'
  * 5 dimensions scored on a 5-Likert scale and visual analogue scale (0 to 100)
  * Higher score means a better outcome
Patient specific questionnaire | T1: baseline (within one week before randomisation)
  Self-administered questions about: gender, ethnicity, age, nationality, weight, height, civil state, mutuality, educational level, year of the breast cancer diagnosis, received breast cancer treatments, lymphedema, medication, other treatments, menopausal, hot flashes.

CONTACTS AND LOCATIONS:
Overall Officials: Jo Nijs, Prof., Principal Investigator — Vrije Universiteit Brussel
Locations (1):
- Vrije Universiteit Brussel (VUB), Jette, Brussels Capital, Belgium

IPD SHARING:
Plan to Share IPD: No